CLINICAL TRIAL: NCT03398317
Title: PICSI vs. MACS for Abnormal Sperm DNA Fragmentation ICSI Cases: a Prospective Randomized Trial
Brief Title: Sperm Selection by Either PICSI or MACS in Cases With Abnormal Sperm DNA Fragmentation Index for ICSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ganin Fertility Center (Other)
Collaborators: The Cleveland Clinic (Other); University of the Western Cape (Other)
Responsible Party: Principal Investigator, Eman Hasanen, Clinical Embryologist, Ganin Fertility Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFC - 002
Record Dates: First submitted 2018-01-07; First posted 2018-01-12 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Sperm DNA Fragmentation
Keywords: SDF; DFI; sperm selection; PICSI; MACS

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICSI (Experimental): Semen processing is done by double layer density gradient method followed by adding Sperm to the dot of hyaluronan on the PICSI dish, within minutes the bound sperm are attached by their acrosome to the surface of the dot. Selecting an individual bound sperm with enhanced genetic and developmental integrity ensures that the sperm selected is the optimal sperm from the sample for oocyte injection
  Interventions: Other: PICSI
- MACS (Active Comparator): Semen processing is done by double layer density gradient method. The resulted pellet is labeled with annexin V microbeads followed by separation on MACS Column, the eluted fraction contains non apoptotic sperm suitable for Oocyte injection.
  Interventions: Other: MACS

INTERVENTIONS:
Other: PICSI — sperm selection using PICSI dish for selecting sperm with lower DNA fragmentation index
  Arms: PICSI
Other: MACS — sperm selection using MACS for selecting sperm with lower DNA fragmentation index
  Arms: MACS

SUMMARY:
On the day of ICSI, choosing the best sperm by either PICSI or magnetic activated cell sorting (MACS) in cases with abnormal DNA is not fully investigated. This study helps in solving this problem by using two known techniques to achieve that purpose.

DETAILED DESCRIPTION:
Sperm DNA fragmentation has shown a negative correlation with fertilization rate, embryo quality, and implantation rate. And a positive correlation with miscarriage rate in the 1st trimester.

Sperm selection methods like PICSI and MACS have been developed for selecting a healthy mature non apoptotic sperm with healthy membrane for Oocyte injection so as to obtain best embryo quality and achieve higher ongoing pregnancy rates.

A sperm selection technique based on sperm membrane binding to hyaluronic acid (PICSI Dish), the main substrate of the oocyte zonapellucida, could improve the likelihood of obtaining better sperm for ICSI with non fragmented DNA. Another sperm selection technique based on Magnetic activated cell sorting (MACS) that depends on the binding of protein Annexin V to phosphatidylserine which is a marker for apoptosis, giving a resulting (eluted) spermatozoa without DNA fragmentation.

In order to determine which sperm selection technique is better for dealing with DNA fragmentation patients we need to study both techniques on two different groups of patients

ELIGIBILITY:
Inclusion Criteria:

* Males diagnosed of abnormal DNA fragmentation index ( > 19%).
* Males with mild to moderate OTA (oligoteratoasthenozoospermia).
* Male aged 18-60 years.
* Female aged 18-40 years.
* Normo responder ( > 5 mature oocytes)
* Male will have to refrain from ejaculation no less than 1 day but no greater than 3 days prior semen specimen production on day of oocyte retrieval

Exclusion Criteria:

Males with normalDNA fragmentation index (<19%)at the initial assessment.

* Leukocytospermia
* Presence of varicocele.
* Known genetic abnormality
* Use of sperm donation or cryopreserved sperm
* Use of Oocyte donation
* Use of gestational carrier
* Presence of any of the endometrial factors that affect embryo implantation such as hydrosalpings, adenomyosis or previous uterine infection
* Any contradictions to undergoing in vitro fertilization or gonadotropin stimulation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 396 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 20 weeks of gestation
  Defined as the proportion of pregnancies that completed more than 20 weeks of gestation

SECONDARY OUTCOMES:
Comparison of cleavage rate | 3 days
  Defined as the proportion of cleaved embryos on day 3 over the injected oocytes
Comparison of Blastulation rate | 5-6 days
  Defined as the proportion of blastocysts formed on day 5 or 6 over the cleaved embryos on day 3
Comparison of Blastocyst quality rate | 5-6 days
  Defined as the assessment of blastocyst quality according to Gardner's criteria into: good, fair or bad in terms of percentage of the total formed blastocysts
Comparison of Pregnancy rate | 14 days following embryo transfer
  Defined as clinical pregnancy per transfer
Comparison of implantation rate | 6- 8 weeks following embryo transfer
  Defined as number of gestational sacs with fetal heart beat, shown by ultrasound in gestational week 6 over number of embryo transferred.

CONTACTS AND LOCATIONS:
Overall Officials: Hosam Zaki, MSc, FRCOG, Study Chair — Ganin Fertility Center, Cairo, Egypt; Eman Hasanen, BSc, Principal Investigator — Ganin Fertility Center, Cairo, Egypt; Khaled El Qusi, BSc, Principal Investigator — Ganin Fertility Center, Cairo, Egypt; Abd El Ghafar Hussin, BSc, Principal Investigator — Ganin Fertility Center, Cairo, Egypt; Salma El Tanbouly, BSc, Principal Investigator — Ganin Fertility Center, Cairo, Egypt; Ashok Agarwal, PhD, Study Director — American Center of Reproductive Medicine, Cleveland Clinic; Ralph Henkel, PhD, Principal Investigator — University of the Western Cape; Hanaa Alkhader, Principal Investigator — Ganin Fertility Center, Cairo, Egypt
Locations (1):
- Ganin Fertility Center, Cairo, Egypt

REFERENCES:
- [Background] Benchaib M, Braun V, Lornage J, Hadj S, Salle B, Lejeune H, Guerin JF. Sperm DNA fragmentation decreases the pregnancy rate in an assisted reproductive technique. Hum Reprod. 2003 May;18(5):1023-8. doi: 10.1093/humrep/deg228. PMID 12721180
- [Background] Baldi and Muratori (2013) Genitic Damage in Human Spermatozoa. USA, NY : Springer Science & Business Media.
- [Derived] Hasanen E, Elqusi K, ElTanbouly S, Hussin AE, AlKhadr H, Zaki H, Henkel R, Agarwal A. PICSI vs. MACS for abnormal sperm DNA fragmentation ICSI cases: a prospective randomized trial. J Assist Reprod Genet. 2020 Oct;37(10):2605-2613. doi: 10.1007/s10815-020-01913-4. Epub 2020 Aug 8. PMID 32772268